CLINICAL TRIAL: NCT00970996
Title: Phase I Biochemotherapy With Cisplatin, Temozolomide, With Increasing Doses of Abraxane, Combined With Interleukin-2 and Interferon in Patients With Metastatic Melanoma
Brief Title: Cisplatin, Temozolomide, Abraxane, With Interleukin-2 and Interferon for Metastatic Melanoma
Acronym: BCAA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0124
Record Dates: First submitted 2009-09-02; First posted 2009-09-03 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-12

CONDITIONS: Melanoma
Keywords: Melanoma; Abraxane; Nab-paclitaxel; Paclitaxel (protein-bound); ABI-007; Cisplatin; Platinol-AQ; Platinol; CDDP; Interleukin 2; IL-2; Proleukin; Intron A; Interferon alpha 2b; Interferon alfa-2b; Temodar; Temozolomide
MeSH Terms: conditions — Melanoma | interventions — Temozolomide; Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel; Taxes; Cisplatin; Interleukin-2; aldesleukin; Interferon alpha-2; Introns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Biochemotherapy (Experimental): Abraxane with Cisplatin, Temozolomide, interleukin-2 and interferon a2b
  Interventions: Drug: Temozolomide; Drug: Abraxane; Drug: Cisplatin; Biological: Interleukin-2; Biological: Interferon alpha 2b

INTERVENTIONS:
Drug: Temozolomide — 250 mg/m^2 by mouth on days 1, 2, and 3 of each 21-day cycle.
  Other Names: Temodar
Drug: Abraxane — 100 mg/m^2 given in a short intravenous infusion 1 hour after completion of Temozolomide and a 2nd dose of 70 mg/m^2 given on day 5 of each 21-day cycle.
  Other Names: Nab-paclitaxel; Paclitaxel (protein-bound); ABI-007
Drug: Cisplatin — 20 mg/m^2 intravenously on days 1, 2, 3, and 4 delivered immediately after Abraxane of each 21-day cycle.
  Other Names: Platinol-AQ; Platinol; CDDP
Biological: Interleukin-2 — 9 MIU/m^2 in a continuous intravenous infusion over 24 hours on days 1, 2, 3, and 4 (total of 96 hours) beginning after completion of Cisplatin of each 21-day cycle.
  Other Names: IL-2; Proleukin
Biological: Interferon alpha 2b — 5 MIU/m^2 in subcutaneous injection on days 1, 2, 3, 4, and 5 of each 21-day cycle.
  Other Names: Intron A

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of Abraxane (nab-paclitaxel) when given in combination with cisplatin, Temodar (temozolomide), interferon alfa-2b, and interleukin-2 (IL-2) to patients with metastatic melanoma.

Primary Objective:

* The primary objective of the Phase I is to determine the toxicity, safety and the maximum tolerated dose maximum tolerated dose of Abraxane in combination with Cisplatin, Temozolomide, interleukin-2 and interferon a2b in patients with metastatic melanoma.

Secondary Objectives:

* To assess responses to the combination.
* To evaluate the duration of response and the overall survival.
* To determine the effectiveness in delaying the appearance of Central Nervous System disease.

DETAILED DESCRIPTION:
The Study Drugs:

Cisplatin, nab-paclitaxel, and temozolomide are chemotherapy drugs and have a direct effect on melanoma cells. Interferon alfa-2b and IL-2 are biotherapy drugs that stimulate the immune system to fight against melanoma. The combination of chemotherapy and biotherapy drugs is called biochemotherapy.

This is the first study using these drugs in combination.

Catheter:

If you are found to be eligible to take part in this study, you will have a central venous catheter (CVC) inserted, if you do not already have one. The catheter is passed through the veins of your arm or the veins that run under your collar bone to reach a wide central vein in the chest that runs above your heart. You will receive a separate consent form for this procedure, which describes the risks.

Nab-paclitaxel, cisplatin, and interleukin-2 are given through this catheter. In certain situations, blood can also be drawn from this catheter.

Study Drug Dose Levels:

You will be assigned to a dose level of nab-paclitaxel based on when you joined this study. Up to 3 dose levels of nab-paclitaxel will be tested. Up to 6 participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of nab-paclitaxel that can be given in combination with the other drugs is found.

All participants will receive the same dose level of temozolomide, cisplatin, interferon alfa-2b, and IL-2.

Study Drug Administration:

Each study cycle will last 3-5 weeks. The length of each cycle will depend on your recovery from the study drugs.

On Day 1 of each cycle:

* You will take temozolomide by mouth.
* You will receive nab-paclitaxel over about 30 minutes by vein about 1 hour after you take temozolomide.
* You will then receive cisplatin by vein. Each infusion of cisplatin will take about 45-120 minutes.
* You will receive interferon alfa-2b by injection into fatty tissue.
* You will begin your IL-2 infusion. The infusion will begin after you receive cisplatin and will continue non-stop until Day 5.

On Day 2 of each cycle:

* You will take temozolomide by mouth.
* You will receive cisplatin by vein about 1 hour after you take temozolomide.
* You will receive interferon alfa-2b by injection into fatty tissue.

On Day 3 of each cycle:

* You will take temozolomide by mouth.
* You will receive cisplatin by vein about 1 hour after you take temozolomide.
* You will receive interferon alfa-2b by injection into fatty tissue.
* Blood (up to 4 teaspoons total) will be drawn for routine tests and tests to check for infection in the blood.

On Day 4 of each cycle:

* You will receive cisplatin by vein.
* You will receive interferon alfa-2b by injection into fatty tissue.
* Blood (up to 4 teaspoons) will be drawn for routine tests.

On Day 5 of each cycle:

* You will receive nab-paclitaxel by vein over about 30 minutes.
* You will receive interferon alfa-2b by injection into fatty tissue.
* Blood (up to 4 teaspoons) will be drawn for routine tests.

Depending on how your body reacts to the study drugs, you will stay in the hospital for 7 or more days.

After you are discharged from the hospital, blood (up to 4 teaspoons) will be drawn 2 times a week for routine tests.

Study Visits:

Before starting each cycle of treatment:

* Your medical history will be recorded.
* You will have a physical exam.
* Blood (about 1-2 tablespoons) will be drawn for routine tests and to check your blood counts.
* You will have a chest x-ray.

After every 2 cycles of treatment, you will have CT scans and an MRI scan of the brain to check the status of the disease. If you have disease in the bone, you will have a PET/CT to check the status of the disease.

If you have skin lesions, you will have them photographed to check the status of the disease.

Length of Study:

You may receive up to 6 cycles of the study drugs. You will be taken off study early if the disease gets worse or intolerable side effects occur.

Follow-Up Contact:

If you are having follow-up visits with a doctor who is not at M. D. Anderson, you will be called 2-4 times a year to learn what treatments you may be receiving and how are you doing. You will continue to receive these calls for as long as possible. The phone calls will take about 5 minutes.

This is an investigational study. Nab-paclitaxel is FDA approved and commercially available for breast cancer. Temozolomide is FDA approved and commercially available for brain cancer. Cisplatin is FDA approved and commercially available for testicular, ovarian, and bladder cancers. Interferon is FDA approved and commercially available for patients with melanoma who are having surgery. IL-2 is FDA approved and commercially available for melanoma and kidney cancer. The combination of these drugs is investigational.

Up to 24 patients will be take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically documented diagnosis of advanced stage IV or unresectable stage III melanoma are eligible.
2. They should have recurrent melanoma with measurable or evaluable sites of disease, 1.0 cm or larger, in order to assess the response to treatment by RECIST.
3. They should not have been exposed to any previous chemotherapy or isolation perfusion for malignant melanoma and have had no previous exposure to interleukin-2. Prior adjuvant interferon is permitted.Prior radiation therapy for metastatic melanoma is permitted provided the patient has un-irradiated metastatic sites for response evaluation and has fully recovered from its toxicity.
4. Patients between 18 years of age and 65 years of age with an expected survival greater than 8 weeks and a Karnofsky performance status of 50% or better or an ECOG performance status of 0, 1 or 2 will be eligible.
5. They should have normal blood counts with a WBC count of more than or equal to 3000/mm^3 an absolute neutrophil count of more than or equal to 1500/mm^3 and a platelet count of more than 100,000/mm^3 and have no impairment of renal function (serum creatinine less than 1.1 mg/dl for females and less than 1.4 mg/dl for males), hepatic function (serum bilirubin level of less than 1.2 mg/dl) and no evidence of significant cardiac or pulmonary dysfunction.
6. They should have no significant intercurrent illness such as an active infection, uncontrolled psychiatric illness, hypercalcemia (calcium greater than 11 mg), or active GI bleeding.

Exclusion Criteria:

1. Patients with bone metastases only.
2. Patients with brain metastases unless their disease has been resected and they are off corticosteroids. Patients with spinal cord compression and leptomeningeal disease. No major surgery or radiation therapy within 21 days before starting treatment.
3. Patients with significant cardiac illness such as symptomatic coronary artery disease or previous history of myocardial infarction, impaired left ventricle function (EF less than 55%) on account of any organic disease such as hypertension or valvular heart disease or serious cardiac arrhythmia requiring therapy. Patients with an EKG disclosing an absolute QT interval greater than 460 msec in the presence of serum potassium greater than or equal 4.0 mEq/L and magnesium greater than/=1.8 mg/dL.
4. Patients with significant impairment of pulmonary function on account of chronic bronchitis or chronic obstructive pulmonary disease (COPD) which has resulted in impairment of vital capacity of FEV1 to less than 75% of predicted normal values.
5. Patients with symptomatic effusions on account of pleural, pericardial or peritoneal metastases of melanoma.
6. Patients who are unable to stay in Houston to receive therapy (first cycle) and/or unable to return for follow-up visits as required by this study.
7. Patients with a history of second malignant tumor, other than the common skin cancers - basal and squamous carcinomas, within the past 5 years and uncertainty about the histological nature of the metastatic lesions.
8. Patients with history of DVT or PE are excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Response Rate | Radiographic studies (CT, MRI scans) to assess disease response after every two cycles (one cycle=21 days).

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas E. Papadopoulos, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T. M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: U.T. M.D. Anderson Cancer Center web page — http://www.mdanderson.org